CLINICAL TRIAL: NCT04291677
Title: Music in Vein in the Intensive Care Unit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Juan Carlos Montejo González (Other)
Responsible Party: Sponsor-Investigator, Juan Carlos Montejo González, Head of Intensive Care Medicine Service, MD, PhD, Hospital Universitario 12 de Octubre
Organization: Hospital Universitario 12 de Octubre (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MUSICALCARE-ICU
Record Dates: First submitted 2020-02-19; First posted 2020-03-02 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Mechanical Ventilation
Keywords: Critical patient; Intensive care unit; Mechanical ventilation; Sedative and analgesic medication; Anxiety; Live musical intervention
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group in which musical intervention (Experimental): Group A: Experimental group in which musical intervention will be applied between the first and the third day of mechanical ventilation.
  Interventions: Other: intervention musical
- Control group (Other): Group B: Control group with standard treatment without musical intervention.
  Interventions: Other: Without intervention musical

INTERVENTIONS:
Other: intervention musical — Intervention group in which musical intervention will be applied the first or third day of mechanical ventilation.
  Arms: Intervention group in which musical intervention
Other: Without intervention musical — Control group with standard treatment without musical intervention.
  Arms: Control group

SUMMARY:
Patients admitted to the Intensive Care Units (ICU) that receive mechanical ventilation need high dose sedative and analgesic medication that may have side effects. Despite this, many of them also experience anxiety and added stress.

Musical intervention is a useful non-pharmacological tool without adverse effects safe and easy to provide for patients with mechanical ventilation admitted to the Intensive Care Units. Its use reduces the use and dose of sedatives, reduces stress and environmental noise. It should be considered in the measures of control of anxiety and noise in the ICU.

The objective of the study is to analyze whether the implementation of a musical intervention can be an effective non-pharmacological intervention in the therapy of patients undergoing mechanical ventilation admitted to an Intensive Care Unit of a High Complexity Hospital.

DETAILED DESCRIPTION:
This is a prospective, randomized clinical study will be developed in the three Units of Intensive Care of the Intensive Medicine Service of the 12 de Octubre Universitarian Hospital. All adult patients admitted to the ICU with requirements for mechanical ventilation and in which the unit's pseudoanalgesia protocol is implemented and having signed your legal representative informed consent to participate in the study will be included. The Patients admitted to the ICU with predictable survival less than 48 hours; those who are not submitted to mechanical ventilation and those whose Legal representative refuses to sign the informed consent wouldn't participate.

The patients will be randomized in two groups: Group A: Intervention group in which musical intervention will be applied between the first and the third day of mechanical ventilation. Group B: Control group with standard treatment without musical intervention.

Live music will be applied every day of the week by professional musicians of the non-profit association Music in Vena (MeV) until mechanical ventilation is removed. There will be sessions of 30 minutes a day. The execution time will be from 13-13:30 hours, and the family will be allowed to participate. The type of music will be classical to be determined by musicians.

The participants will be followed for the duration invasive mechanical ventilation.

The Investigators of this project ensure that the principalities ethics for medical research in beings humans of the HELSINKI DECLARATION OF THE WORLD MEDICAL ASSOCIATION have been adapted. MUSICALCARE-ICU has been approved by the Ethics Committee of the 12 de Octubre Universitarian Hospital. The legal representative must give written informed consent to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted to the ICU with requirements for mechanical ventilation and in which the unit's pseudoanalgesia protocol is implemented.
* A legal representative informed consent to participate in the study has to be signed.

Exclusion Criteria:

* Patients admitted to the ICU with predictable survival less than 48 hours.
* Patients who are not subjected to mechanical ventilation.
* Patients whose Legal representative refuses to sign the informed consent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Total and extra pseudoanalgesia requirements change. | It will be analyzed at baseline, at the end of the musical intervention, at 30 minutes, 60 minutes and at 8 hours after the intervention.
  Change of the anxiety and pain level in patients with invasive mechanical ventilation with music therapy.

SECONDARY OUTCOMES:
Change of Heart rate. | It will be analyzed at baseline, at the end of the musical intervention, at 30 minutes, 60 minutes and at 8 hours after the intervention.
  Change of the heart rate registered in electrocardiogram in patients with invasive mechanical ventilation with music therapy.
Change of systolic blood pressure; diastolic blood pressure and mean blood pressure. | It will be analyzed at baseline, at the end of the musical intervention, at 30 minutes, 60 minutes and at 8 hours after the intervention.
  Change systolic blood pressure; diastolic blood pressure and average blood pressure.
Change vasoactive drug requirements. | It will be analyzed at baseline, at the end of the musical intervention, at 30 minutes, 60 minutes and at 8 hours after the intervention.
  Percentage of patients who experience a change of the vasoactive drug requirements in patients with invasive mechanical ventilation with music therapy.
Blood glucose control. | It will be analyzed at baseline, at the end of the musical intervention, at 30 minutes, 60 minutes and at 8 hours after the intervention.
  Percentage of patients who normalize blood glucose levels (range 70-110 milligrams/deciliter).
Change insulin requirements. | It will be analyzed at baseline, at the end of the musical intervention, at 30 minutes, 60 minutes and at 8 hours after the intervention.
  Percentage of patients who change insulin requirements measured as International Unit per day (IU/day).
Change cortisol and growth hormone level. | It will be performed at 9 hours, prior to the implementation of the musical intervention, and at 30 minutes after the end of the intervention on days 1, 3, 7 and 10.
  Change serum levels biomarkers (cortisol and growth hormone level) in patients with invasive mechanical ventilation with music therapy.
Change the stay in the Intensive Care Unit (ICU) | At 90 days
  Change in mechanical ventilation time in patients with musical intervention reduces ICU stay.
Quality of Life (HRQoL) according to Karnofsky's index. | At 90 days
  Change in the Quality of Life (QoL) will be measured using the Karnofsky Performance Status other method to assess the functional status of a patient. The Karnofsky index, between 100 and 0.
  100-Normal, no complaints; no evidence of disease. 90-Able to carry on normal activity; minor signs or symptoms of disease. 80-Normal activity with effort, some signs or symptoms of disease. 70-Cares for self but unable to carry on normal activity or to do active work. 60-Requires occasional assistance but is able to care for most of personal needs.
  50-Requires considerable assistance and frequent medical care. 40-Disabled; requires special care and assistance. 30-Severely disabled; hospitalization is indicated although death not imminent. 20-Very ill; hospitalization and active supportive care necessary. 10-Moribund 0-Dead
The overall Health related Quality of Life (HRQoL) of patients with requirements for mechanical ventilation will be measured using a patient self rating questionnaire. | At 90 days
  Change in the Quality of Life (QoL) will be measured using the Eastern Cooperative Oncology Group (ECOG) Scale of Performance Status who describes a patient's level of functioning in terms of their ability to care for themselves, daily activity, and physical ability (walking, working, etc.).
  Grade 0: Fully active, able to carry on all pre-disease performance without restriction.
  Grade 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  Grade 2: Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours.
  Grade 3: Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours Grade 4: Completely disabled; cannot carry on any selfcare; totally confined to bed or chair Grade 5: Dead.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Carlos Montejo, PhD MD, Study Chair — Hospital Universitario 12 de Octubre
Locations (1):
- Hospital Universitario 12 de Octubre, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No